CLINICAL TRIAL: NCT02910037
Title: Clinical Implementation of Metagenomic Next-Generation Sequencing for Precision Diagnosis of Acute Infectious Diseases; Neuroinflammatory Cohort
Brief Title: Precision Diagnosis of Acute Infectious Diseases; Neuroinflammatory Cohort
Acronym: PDAID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: California Initiative to Advance Precision Medicine (Other); Sandler Foundation (Unknown); Bowes Foundation (Unknown); Charles and Helen Schwab Foundation (Unknown); University of California, Davis (Other); University of California, Los Angeles (Other); Children's Hospital Los Angeles (Other); Children's Hospital Colorado (Other); St. Jude Children's Research Hospital (Other); Children's National Research Institute (Other); University of California, Berkeley (Other); DNAnexus, Inc. (Unknown); Syapse, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P0509948
Record Dates: First submitted 2016-09-13; First posted 2016-09-21 (Estimated); Results first posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Encephalitis; Meningitis
Keywords: metagenomic next-generation sequencing; microbiological diagnosis; bacterial infections; viral infections; fungal infections; parasitic infections
MeSH Terms: conditions — Encephalitis; Meningitis; Bacterial Infections; Virus Diseases; Mycoses; Parasitic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- patients enrolled for mNGS testing (Experimental): Patients with meningitis and/or encephalitis will be enrolled in this study in order to analyze the clinical utility of mNGS for pathogen detection. There is no control group for this study (Investigators will identify historical controls by retrospective chart review and clinical reimbursement documents).
  Interventions: Device: mNGS for pathogen detection

INTERVENTIONS:
Device: mNGS for pathogen detection — This assay is a laboratory-validated metagenomic test for comprehensive detection of viruses, bacteria, fungi, and parasites in clinical samples.
  Other Names: Sequence-Based Ultrarapid Pathogen Identification (SURPI)+; UCSF metagenomic next-generation sequencing testing

SUMMARY:
This study aims to use a clinically validated metagenomic next-generation sequencing (mNGS) assay to provide a demonstration of precision medicine for diagnosis of acute infectious disease in hospitalized patients. From June 2016 to June 2017, 200 patients will be enrolled from multiple hospitals in California and outside of California. Patients will be evaluated to determine the impact on the mNGS assay on diagnostic yield, hospital costs and clinical outcomes.

DETAILED DESCRIPTION:
This study aims to use a clinically validated metagenomic next-generation sequencing (mNGS) assay to provide a demonstration of precision medicine for diagnosis of acute infectious disease in hospitalized patients, with the goal of directly impacting clinical care and improving patient mortality. This diagnostic test has been previously validated in a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory, the University of California, San Francisco Clinical Microbiology Laboratory. From June 2016 to June 2017, investigators will prospectively enroll 200 patients from multiple hospitals in California (University of California, San Francisco; University of California, Los Angeles; University of California, Davis; Children's Hospital Los Angeles) and outside California (Children's National Medical Center, Children's Hospital Colorado, St. Jude Children's Research Hospital) for mNGS testing, and evaluate the impact on the assay on diagnostic yield, hospital costs and clinical outcomes.

ELIGIBILITY:
Exclusions:

* Patients on a 5150 or 5250 psychiatric hold
* Prisoners
* University of California employees / students or close associates of any of the key personnel on the study
* Outpatients and/or patients with chronic illness

Inclusion:

Demographic Criteria

1. Age: any (no age limit)
2. Language: any (with the use of interpreting services for obtaining consent)

For the following, the infectious syndromes include meningitis, encephalitis, fever, sepsis, and pneumonia:

Clinical Criteria

1. Hospital admission or transfer with diagnosis of an presumed infectious syndrome or clinical presentation consisting with an infectious syndrome, as defined below:

   * Meningitis: fever >38°C and abnormal imaging or CSF pleocytosis (CSF white blood cell count (WBC) > 5 /mm^3) +/- stiff neck, +/- headache, +/- seizure
   * Encephalitis: pleocytosis and at least one of the following: altered mental status, seizures, new onset of focal neurologic findings, abnormal EEG, acute brain abnormalities on neuroimaging
2. No known diagnosis of non-infectious etiology responsible for symptoms
3. Time of enrollment: within 7 days of onset of symptoms, either initial presentation or acute exacerbation of presumed infectious syndrome.

Specimen Criteria

1. cerebrospinal fluid available within 7 days of symptom onset AND within 3 days of hospital admission or transfer unless evidence for acute exacerbation as defined by abrupt decline in clinical status, worsening pleocytosis or other laboratory parameters
2. Minimum of 600 microliters (uL) of clinical sample, stored at 4 degrees Celsius (C) no more than 5 days (ideally frozen in -70 degrees Celsius within 24 hours of collection)
3. No more than 3 freeze-thaw cycles

Ages: 1 Minute to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Y Chiu, MD, PhD, Principal Investigator — University of California, San Francisco; Hannah Sample, BS, Study Director — University of California, San Francisco
Locations (7):
- United States (7):
  - University of California, Davis Medical Center, Davis, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California, Los Angeles Medical Center, Los Angeles, California
  - University of California, San Francisco Medical Center, San Francisco, California
  - Children's Hospital Colordao, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - St. Jude Children's Research Hospital, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
All genomic / metagenomic sequencing data from this study will be made available either at NIH Sequence Read Archive or NIH database of Genotypes and Phenotypes (dbGaP), depending on whether human sequence data is included. The investigators intend to make de-identified ancillary clinical, laboratory, and radiographic data available as well upon request.
Supporting Information: CSR
Time Frame: The clinical study report will be submitted for publication by June 2018.
URL: http://nextgendiagnostics.ucsf.edu/our-research/

REFERENCES:
- [Background] Wilson MR, Naccache SN, Samayoa E, Biagtan M, Bashir H, Yu G, Salamat SM, Somasekar S, Federman S, Miller S, Sokolic R, Garabedian E, Candotti F, Buckley RH, Reed KD, Meyer TL, Seroogy CM, Galloway R, Henderson SL, Gern JE, DeRisi JL, Chiu CY. Actionable diagnosis of neuroleptospirosis by next-generation sequencing. N Engl J Med. 2014 Jun 19;370(25):2408-17. doi: 10.1056/NEJMoa1401268. Epub 2014 Jun 4. PMID 24896819
- [Background] Greninger AL, Messacar K, Dunnebacke T, Naccache SN, Federman S, Bouquet J, Mirsky D, Nomura Y, Yagi S, Glaser C, Vollmer M, Press CA, Kleinschmidt-DeMasters BK, Dominguez SR, Chiu CY. Clinical metagenomic identification of Balamuthia mandrillaris encephalitis and assembly of the draft genome: the continuing case for reference genome sequencing. Genome Med. 2015 Dec 1;7:113. doi: 10.1186/s13073-015-0235-2. PMID 26620704
- [Background] Naccache SN, Peggs KS, Mattes FM, Phadke R, Garson JA, Grant P, Samayoa E, Federman S, Miller S, Lunn MP, Gant V, Chiu CY. Diagnosis of neuroinvasive astrovirus infection in an immunocompromised adult with encephalitis by unbiased next-generation sequencing. Clin Infect Dis. 2015 Mar 15;60(6):919-23. doi: 10.1093/cid/ciu912. Epub 2015 Jan 7. PMID 25572898
- [Background] Greninger AL, Naccache SN, Messacar K, Clayton A, Yu G, Somasekar S, Federman S, Stryke D, Anderson C, Yagi S, Messenger S, Wadford D, Xia D, Watt JP, Van Haren K, Dominguez SR, Glaser C, Aldrovandi G, Chiu CY. A novel outbreak enterovirus D68 strain associated with acute flaccid myelitis cases in the USA (2012-14): a retrospective cohort study. Lancet Infect Dis. 2015 Jun;15(6):671-82. doi: 10.1016/S1473-3099(15)70093-9. Epub 2015 Mar 31. PMID 25837569
- [Background] Naccache SN, Federman S, Veeraraghavan N, Zaharia M, Lee D, Samayoa E, Bouquet J, Greninger AL, Luk KC, Enge B, Wadford DA, Messenger SL, Genrich GL, Pellegrino K, Grard G, Leroy E, Schneider BS, Fair JN, Martinez MA, Isa P, Crump JA, DeRisi JL, Sittler T, Hackett J Jr, Miller S, Chiu CY. A cloud-compatible bioinformatics pipeline for ultrarapid pathogen identification from next-generation sequencing of clinical samples. Genome Res. 2014 Jul;24(7):1180-92. doi: 10.1101/gr.171934.113. Epub 2014 Jun 4. PMID 24899342
- [Background] Wilson MR, Shanbhag NM, Reid MJ, Singhal NS, Gelfand JM, Sample HA, Benkli B, O'Donovan BD, Ali IK, Keating MK, Dunnebacke TH, Wood MD, Bollen A, DeRisi JL. Diagnosing Balamuthia mandrillaris Encephalitis With Metagenomic Deep Sequencing. Ann Neurol. 2015 Nov;78(5):722-30. doi: 10.1002/ana.24499. Epub 2015 Aug 24. PMID 26290222
- [Result] Wilson MR, Sample HA, Zorn KC, Arevalo S, Yu G, Neuhaus J, Federman S, Stryke D, Briggs B, Langelier C, Berger A, Douglas V, Josephson SA, Chow FC, Fulton BD, DeRisi JL, Gelfand JM, Naccache SN, Bender J, Dien Bard J, Murkey J, Carlson M, Vespa PM, Vijayan T, Allyn PR, Campeau S, Humphries RM, Klausner JD, Ganzon CD, Memar F, Ocampo NA, Zimmermann LL, Cohen SH, Polage CR, DeBiasi RL, Haller B, Dallas R, Maron G, Hayden R, Messacar K, Dominguez SR, Miller S, Chiu CY. Clinical Metagenomic Sequencing for Diagnosis of Meningitis and Encephalitis. N Engl J Med. 2019 Jun 13;380(24):2327-2340. doi: 10.1056/NEJMoa1803396. PMID 31189036
- [Result] Chiu CY, Coffey LL, Murkey J, Symmes K, Sample HA, Wilson MR, Naccache SN, Arevalo S, Somasekar S, Federman S, Stryke D, Vespa P, Schiller G, Messenger S, Humphries R, Miller S, Klausner JD. Diagnosis of Fatal Human Case of St. Louis Encephalitis Virus Infection by Metagenomic Sequencing, California, 2016. Emerg Infect Dis. 2017 Oct;23(10):1964-1968. doi: 10.3201/eid2310.161986. PMID 28930022
- [Result] Murkey JA, Chew KW, Carlson M, Shannon CL, Sirohi D, Sample HA, Wilson MR, Vespa P, Humphries RM, Miller S, Klausner JD, Chiu CY. Hepatitis E Virus-Associated Meningoencephalitis in a Lung Transplant Recipient Diagnosed by Clinical Metagenomic Sequencing. Open Forum Infect Dis. 2017 Jun 13;4(3):ofx121. doi: 10.1093/ofid/ofx121. eCollection 2017 Summer. PMID 28721353
- See also: brief description of PDAID study and referral link — http://chiulab.ucsf.edu
- See also: summary of the PDAID project, sponsored by the California Initiative to Advance Precision Medicine — http://www.ciapm.org/project/precision-diagnosis-acute-infectious-diseases
- See also: video describing metagenomic next-generation sequencing and its use for diagnosis of infections — https://www.youtube.com/watch?v=OFYSEowGfeI
- See also: The UCSF Center for Next-Gen Precision Diagnostics — http://nextgendiagnostics.ucsf.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Enrolled for mNGS Testing
Started | 214
Completed | 204
Not Completed | 10
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | Patients Enrolled for mNGS Testing
Number analyzed (Participants) | 204
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 45
  Between 18 and 65 years | 124
  >=65 years | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (22.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 114
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 17
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 118
  More than one race | 42
  Unknown or Not Reported | 13
Region of Enrollment [Number; unit: participants]
  United States | 204

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Cases With at Least One Provider Response
Description: Investigators will evaluate impact of mNGS assay by clinician surveys and Clinical Microbial Sequencing Board (CMSB) feedback and discussion as measured by at least 1 provider response per case.
Time Frame: within 1 month of patient enrollment in study
Population: Treating teams for 204 included patients
Measure: Number; unit: cases
Groups:
- Pre mNGS Result Feedback From Providers: Response from treating clinicians regarding differential for patients before mNGS for pathogen detection was resulted.
- Post mNGS Results Feedback From Providers: Response for survey from treating clinicians regarding differential and impact of mNGS results on care.
Arm/Group | Pre mNGS Result Feedback From Providers | Post mNGS Results Feedback From Providers
Number analyzed (Participants) | 204 | 204
cases | 98 | 58

2. Secondary Outcome: Clinical Outcomes: Time From Cerebrospinal Fluid Collection to mNGS Results
Description: Investigators will review medical records to determine time of initial presentation and measure the time to mNGS results.
Time Frame: from admission to 1 month post discharge for each patient during the enrollment period of study
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Patients Enrolled for mNGS Testing
Number analyzed (Participants) | 204
days | 13.5 (4.8)

3. Secondary Outcome: Clinical Outcomes: Length of Stay
Description: Investigators will review medical records to determine length of stay including discharge to rehab facilities.
Time Frame: from admission to 1 month post discharge for each patient during the enrollment period of study
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Patients Enrolled for mNGS Testing
Number analyzed (Participants) | 204
days | 27.9 (32.5)

4. Secondary Outcome: Clinical Outcomes: Final Diagnosis Category
Description: Investigators will review medical records to determine final diagnosis after all diagnostic testing has been performed including metagenomic Next-Gen sequencing and autopsy where applicable.
Time Frame: from admission to time of final case review (1 month post discharge or up to one year)
Measure: Count of Participants; unit: Participants
Groups:
- Autoimmune: Patients that received a definitive autoimmune diagnosis for their CNS disease.
- Infectious: Patients that received a definite infectious disease diagnosis for their CNS disease.
- Neoplastic: Patients that received a definitive neoplastic diagnosis for their CNS disease.
- Post Infectious: Patients that received a definitive post infectious diagnosis for their CNS disease.
- Toxic Metabolic: Patients that received a definitive toxic metabolic diagnosis for their CNS disease.
- Structural: Patients that received a definitive structural diagnosis for their CNS disease.
- Vascular: Patients that received a definitive vascular diagnosis for their CNS disease.
- Other: Patients that received a definitive diagnosis for their CNS disease in another category.
- Unknown: Patients that did not received a definitive diagnosis for their CNS disease.
Arm/Group | Autoimmune | Infectious | Neoplastic | Post Infectious | Toxic Metabolic | Structural | Vascular | Other | Unknown
Number analyzed (Participants) | 204 | 204 | 204 | 204 | 204 | 204 | 204 | 204 | 204
Participants | 17 | 57 | 7 | 3 | 3 | 0 | 1 | 15 | 101

5. Secondary Outcome: Clinical Outcomes: Concordance of mNGS With Other Molecular Testing on Cerebrospinal Fluid Pathogens
Description: mNGS findings were compared to conventional testing for concordance. Conventional testing included both tests that were ordered as part of each patients workup and those order to confirm mNGS findings on cerebrospinal fluid (CSF).
Time Frame: from admission to 1 month post discharge for each patient during the enrollment period of study
Measure: Count of Participants; unit: Participants
Groups:
- mNGS Only Diagnosis, Confirmation Attempted: mNGS only diagnosis, confirmation attempted on remnant CSF and/or ancillary specimen(s) (i.e. brain biopsy)
- Concordant With Conventional Testing: mNGS and conventional direct detection testing resulted in the same finding. Direct detection included culture and PCR. Results were considered concordant for this measure if conventional testing was positive by indirect testing (i.e. antibody) and both direct detection (i.e. PCR) and mNGS were negative.
- Missed by mNGS: Missed by mNGS, includes those with reads under established reporting thresholds
- False Positive by mNGS: False positives were reported when mNGS resulted an organism that was not detected by other method (direct and/or indirect) and was not thought to be clinically relevant by the treating clinicians. Incidental findings (i.e. HIV) were not reported as false positives.
- mNGS Only Finding, Unable to Confirm: mNGS only finding, unable to confirm due to test or specimen unavailability
Arm/Group | mNGS Only Diagnosis, Confirmation Attempted | Concordant With Conventional Testing | Missed by mNGS | False Positive by mNGS | mNGS Only Finding, Unable to Confirm
Number analyzed (Participants) | 204 | 204 | 204 | 204 | 204
Participants | 16 | 174 | 9 | 1 | 4

ADVERSE EVENTS:
Time Frame: up to 1.5 years, 30 day mortality is reported
Arm/Group | Patients Enrolled for mNGS Testing
All-Cause Mortality (participants affected / at risk) | 23/204
Serious Adverse Events (participants affected / at risk) | 0/204
Other Adverse Events (participants affected / at risk) | 0/204

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT02910037/Prot_SAP_000.pdf